CLINICAL TRIAL: NCT00626210
Title: Modafinil Treatment for Sleep/Wake Disturbances in Older Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, VA Palo Alto Health Care System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8564
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders; Alzheimer Disease
Keywords: Mild Cognitive Impairment (MCI); Sleep; Fatigue; Memory
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alzheimer Disease; Cognitive Dysfunction; Fatigue | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modafinil (Experimental)
  Interventions: Drug: modafinil

INTERVENTIONS:
Drug: modafinil — 100-400 mg daily for 4 weeks
  Other Names: Provigil

SUMMARY:
Modafinil, trade named Provigil, is a medication approved by the Food and Drug Administration for the treatment of narcolepsy, obstructive sleep apnea/hypopnea syndrome, and shift work sleep disorder. Each of these problems is characterized by difficulty sleeping at night and excessive daytime sleepiness. Modafinil is prescribed during the day to counteract this sleepiness. The idea behind this treatment is that sleepiness that leads to napping during the day prevents a patient from being tired or sleepy enough to get good sleep at night. This study is designed to determine if the medication can "reset" participants' sleep/wake rhythm to a more normal rhythm.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Alzheimer's disease or Mild Cognitive Impairment
* Subjective complaint of sleep disruption, unsatisfactory sleep, early morning awakening, early bedtime, or excessive daytime sleepiness. Such complaint can be made by either the potential participant or by the caregiver.

Exclusion Criteria:

* Participation in any other clinical drug trial
* Liver failure
* Believed by the investigator to be unwilling or unable to follow the protocol
* Active liver or coronary disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zeitzer, PhD, Principal Investigator — Stanford University/VAPAHCS
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Zeitzer JM, Buckmaster CL, Parker KJ, Hauck CM, Lyons DM, Mignot E. Circadian and homeostatic regulation of hypocretin in a primate model: implications for the consolidation of wakefulness. J Neurosci. 2003 Apr 15;23(8):3555-60. doi: 10.1523/JNEUROSCI.23-08-03555.2003. PMID 12716965
- [Background] Wisor JP, Nishino S, Sora I, Uhl GH, Mignot E, Edgar DM. Dopaminergic role in stimulant-induced wakefulness. J Neurosci. 2001 Mar 1;21(5):1787-94. doi: 10.1523/JNEUROSCI.21-05-01787.2001. PMID 11222668
- [Background] Scammell TE, Estabrooke IV, McCarthy MT, Chemelli RM, Yanagisawa M, Miller MS, Saper CB. Hypothalamic arousal regions are activated during modafinil-induced wakefulness. J Neurosci. 2000 Nov 15;20(22):8620-8. doi: 10.1523/JNEUROSCI.20-22-08620.2000. PMID 11069971
- [Background] Lambe EK, Olausson P, Horst NK, Taylor JR, Aghajanian GK. Hypocretin and nicotine excite the same thalamocortical synapses in prefrontal cortex: correlation with improved attention in rat. J Neurosci. 2005 May 25;25(21):5225-9. doi: 10.1523/JNEUROSCI.0719-05.2005. PMID 15917462
- [Background] Saper CB, German DC. Hypothalamic pathology in Alzheimer's disease. Neurosci Lett. 1987 Mar 9;74(3):364-70. doi: 10.1016/0304-3940(87)90325-9. PMID 2436113
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil: daily 100 mg of modafinil within 1 hr of awakening for one week followed by daily 200 mg of modafinil within 1 hr of awakening for one week
Period: Overall Study
Arm/Group | Modafinil
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Modafinil: Open label study in which all participants get modafinil
Arm/Group | Modafinil
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Sleep Length at 1 Month
Time Frame: 1 month
Measure: Median (Full Range); unit: hours
Arm/Group | Modafinil
Number analyzed (Participants) | 2
hours | 9.5 [9.5 to 9.5]

2. Secondary Outcome: Improvement of Daytime Alertness and Quality of Life.
Time Frame: ~1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Modafinil
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes